CLINICAL TRIAL: NCT03347461
Title: Otiprio Versus Ciprodex to Reduce Tympanostomy Tube Failure
Brief Title: Otiprio Versus Ciprodex Tympanostomy Tube Outcomes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Low use of Otiprio among otolaryngologists.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-37078
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Otorrhea; Otitis Media With Effusion in Children
Keywords: Tympanostomy tube placement; Otiprio; Ciprodex drops; Ear drops; Middle ear
MeSH Terms: interventions — Ciprofloxacin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Otiprio by surgeon (Experimental): Otiprio will be administered through the tympanic membrane by the otolaryngologist immediately after tympanostomy placement.
  Interventions: Drug: Otiprio
- Ciprodex by surgeon (Active Comparator): Ciprodex drops will be instilled by the otolaryngologist into the affected ear immediately after tympanostomy surgery.
  Interventions: Drug: Ciprodex
- Ciprodex by surgeon and parent (Active Comparator): Ciprodex drops will be instilled by the otolaryngologist into the ear immediately after tympanostomy tube surgery. The parent or guardian will administer Ciprodex drops into the ears twice daily for five days after surgery.
  Interventions: Drug: Ciprodex

INTERVENTIONS:
Drug: Otiprio — Otiprio is a single-dose, physician-administered, sustained-exposure otic fluoroquinolone antibacterial for the treatment of pediatric patients with bilateral otitis media with effusion undergoing tympanostomy tube placement surgery. Otoprio (6% ciprofloxacin, 60 mg/mL) will be administered through the tube lumen by the otolaryngologist immediately after tympanostomy surgery.
  Other Names: ciprofloxacin otic suspension
  Arms: Otiprio by surgeon
Drug: Ciprodex — Ciprodex is a combined antibiotic and steroid ear drop used to treat otitis media with tympanostomy tubes. Four drops of Ciprodex (0.14mL) instilled by the otolaryngologist into the affected ear immediately after tympanostomy surgery. Each mL of Ciprodex contains ciprofloxacin hydrochloride 0.3 % (equivalent to 3 mg ciprofloxacin base) and dexamethasone 0.1 % equivalent to 1 mg dexamethasone
  Other Names: ciprofloxacin and dexamethasone
  Arms: Ciprodex by surgeon; Ciprodex by surgeon and parent

SUMMARY:
Otolaryngologists routinely administer ear drops at the time of tympanostomy tube placement in order to prevent tube otorrhea; however, there is a lack of consensus as to which drops are the most effective, and whether a post-operative regimen should be used. Utilizing drops postoperatively places the onus of administration on parents who may have various difficulties in delivering the drops to their child's ears. Additionally, prescribing drops postoperatively is a health care cost. The purpose of this study is to determine if there is a difference in prevention of tympanostomy tube failure (defined as tube blockage or otorrhea) between Otiprio administered once intraoperatively, Ciprodex otic dropgs administered once intraoperatively, and Ciprodex otic drops administered intraoperatively with a postoperative course.

DETAILED DESCRIPTION:
Tympanostomy tube placement is indicated in children with recurrent acute otitis media or chronic otitis media with effusion. Ear dishcarge, otorrhea, is the most common complication following tympanostomy tube placement and occurs in up to 25% of patients. Otorrhea can lead to tube obstruction, making the tube ineffective in ventilating the middle ear or improving hearing. Otolaryngologists routinely administer ear drops at the time of tympanostomy tube placement in order to prevent otorrhea and tube blockage; however, there is lack of consensus as to which drops are the most effective and what dosing regimen should be used.

Options for prevention of otorrhea and tympanostomy tube blockage include intraoperative single-dose application of topical drops or postoperative prolonged application of topical drops. One issue with the prolonged application of drops after surgery is the requirement of parents to administer the drops at home. Thus, the delivery of medication to the middle ear is variable given the difficulty of administering ear drops to a child. Another option exists as a one-time application at the time of surgery, but provides an extended duration of medication in the middle ear. Otiprio is a single-dose suspension of ciprofloxacin and has been FDA approved since February 2015 for use in pediatric patients with otitis media with effusion who require tympanostomy tube placement. Otiprio exists as a liquid at or below room temperature and transitions into a gel after exposure to body temperature in the middle ear. Administrated as an injection into the middle ear at the time of tympanostomy tube placement, Otipiro slowly releases antibiotic treatment over the course of a week, eliminating the need for parents to administer drops.

The study is a prospective, randomized (1:1:1), single-blind, trial of three treatment groups in pediatric subjects with bilateral middle ear effusion who require tympanostomy tube placement. Approximately 300 subjects will be randomized: 100 randomized to receive Otiprio intraoperatively, 100 randomized to receive Ciprodex intraoperatively, and 100 randomized to receive Ciprodex intraoperatively with five days of Ciprodex drops postoperatively.

All participants will undergo tympanostomy tube placement in the operating room as clinically indicated by an Otolaryngologist. Prior to the surgery, the patient will be randomized to one of the three trial arms. During the operation, the surgeon, who will be blinded until completion of tube placement as to which arm the participant is randomized, will administer Otiprio as a one-time intratympanic injection or Ciprodex, by administering 3-5 drops into each ear canal. For the trial arm that includes a 5 day course of Ciprodex postoperatively, the patient's parents will be instructed on how to administer the drops. As per standard of care, all participants will be assessed at a postoperative visit 2-4 weeks post surgery. A blinded assessor to the randomized study arm will perform otoscopy (ear exam) during that visit to determine if there is presence of otorrhea or tympanostomy tube blockage.

ELIGIBILITY:
Inclusion Criteria:

* Children (6 months to 10 years)
* Clinical diagnosis of bilateral middle ear effusion or recurrent acute otitis media requiring tympanostomy tube placement

Exclusion Criteria:

* Patient having any other concurrent surgery
* History of mastoid surgery, chronic or recurrent bacterial infections
* Tympanic membrane perforations
* History of immunodeficiency disease
* Abnormalities of the tympanic membrane or middle ear
* Otic or systemic corticosteroid within 7 days of surgery
* Topical or systemic antimicrobials or antifungal agents prior to their particular washout intervals
* Concurrent use of anti-inflammatory agents
* Allergy to the medications used in this study and their components
* Menarcheal or postmenarcheal female.

Ages: 6 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Post operative otorrhea | Post operative visit 2-4 weeks after tube placement
  Otorrhea is drainage from the ear. Evaluation will be performed by a blind assessor via otoscopy.
Tympanostomy tube blockage | Post operative visit 2-4 weeks after tube placement
  Tympanostomy tube blockage is when the placed tube becomes clogged or obstructed. Evaluation will be performed by a blind assessor via otoscopy.

SECONDARY OUTCOMES:
Resolution of effusion post operatively | Post operative visit 2-4 weeks after tube placement
  Effusion is the presence of middle ear fluid. Evaluation will be performed by a blind assessor via otoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Weber, MD, Study Chair — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided